CLINICAL TRIAL: NCT07045376
Title: Effects of Multi-strategy Evidence-based Education Training Programs on Knowledge, Attitude, and Preventive Behavior Towards Surgical Smoke Hazards Among Operating Room Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, CHIU-MIN KUO, Principal Investigator, Chang Gung University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202401687B0
Record Dates: First submitted 2025-06-07; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Electrocautery Smoke
Keywords: surgical smoke; evidence-based multi-strategy educational training program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- develop an evidence-based multi-strategy educational training program on surgical smoke (Experimental): Based on evidence from the literature, the content of the evidence-based multi-strategy educational training program includes:
  Providing a surgical smoke protection handbook and displaying environmental education posters.
  Using an official LINE account to disseminate knowledge about surgical smoke, protective techniques, and related information.
  Organizing a hands-on workshop on surgical smoke hazard prevention, allowing participants to practice operating smoke evacuation equipment.
  Interventions: Other: evidence-based multi-strategy educational training program on surgical smoke

INTERVENTIONS:
Other: evidence-based multi-strategy educational training program on surgical smoke — Based on evidence from the literature, the content of the evidence-based multi-strategy educational training program includes:
  Providing a surgical smoke protection handbook and displaying environmental education posters.
  Using an official LINE account to disseminate knowledge about surgical smoke, protective techniques, and related information.
  Organizing a hands-on workshop on surgical smoke hazard prevention, allowing participants to practice operating smoke evacuation equipment.

SUMMARY:
This study aims to: 1) develop an evidence-based multi-strategy educational training program on surgical smoke, and 2) investigate the effectiveness of the "evidence-based multi-strategy educational training program" on operating room nurses' knowledge, attitudes, and preventive behaviors concerning the hazards of surgical smoke.

The research questions of this study are as follows:

What are the levels of knowledge, attitudes, and preventive behaviors regarding surgical smoke hazards among operating room nurses?

What is the effect of an "evidence-based multi-strategy educational training program" on operating room nurses' knowledge of surgical smoke hazards?

What is the effect of an "evidence-based multi-strategy educational training program" on operating room nurses' attitudes toward surgical smoke hazards?

What is the effect of an "evidence-based multi-strategy educational training program" on operating room nurses' preventive behaviors regarding surgical smoke hazards? The experimental group received the "evidence-based multi-strategy educational training program on surgical smoke," while the control group received the conventional training on surgical smoke. Measurements were taken three times: a pretest, a post-test one week after the course, and a follow-up test four weeks later. The research tools included a self-designed questionnaire that included scales on knowledge, attitudes toward surgical smoke, and self-protective behaviors.

DETAILED DESCRIPTION:
To avoid cross-contamination during the research process, participants in the experimental and control groups were recruited from different hospitals. After obtaining approval from administrative supervisors at a regional hospital and a medical center in southern Taiwan, the researcher explained the study purpose and procedures to interested nurses and obtained their informed consent in writing.

1. If you work at Chiayi Chang Gung Memorial Hospital, you will be assigned to the experimental group and will receive a four-week multi-strategy evidence-based educational training program on surgical smoke.
2. If you work at Kaohsiung Chang Gung Memorial Hospital, you will be assigned to the control group and will receive a four-week standard in-service training on surgical smoke provided by the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Operating room nurses who have been formally employed for more than three months.
2. Willing to participate in the study and sign the informed consent form.
3. Possess a mobile phone or computer with internet access. -

Exclusion Criteria:

- Operating room nurses who are in training, internship, part-time student positions, or currently on parental leave.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
This study adopted the Chinese questionnaire developed by Yu et al. (2021) as the data collection tool. the Surgical Smoke Knowledge Scale (17 items),the Attitude Toward Surgical Smoke Scale (11 item)sand the Preventive BehaviorScale (10 items). | one week after the course (post-test) and at the fourth week (follow-up post-test).
  Changes in operating room nurses' knowledge, attitudes, and preventive behaviors regarding surgical smoke hazards will be measured one week after the course (post-test) and at the fourth week (follow-up post-test).

CONTACTS AND LOCATIONS:
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Chang Gung Medical Foundation, Chiayi City, Puzi City, Taiwan

IPD SHARING:
Plan to Share IPD: No